CLINICAL TRIAL: NCT04356885
Title: Impact of Containment and Quarantine During COVID-19 Outbreack on Psychotic Symptoms in the General Population in France
Brief Title: COVID-19 and Psychotic Symptoms in France
Acronym: SCHIZOVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Epsylon Laboratory, EA 4556, University Paul Valéry Montpellier 3, France (Unknown); Laboratoy LIP/PC2S, University Grenobles-Alpes, Grenoble, France (Unknown); Centre référent de réhabilitation psychosociale de Grenoble, Grenoble, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0225
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study the impact of containment related to COVID-19 pandemic on psychotic experiences in the general population in France.

DETAILED DESCRIPTION:
The pandemic of the novel coronavirus disease (COVID-19) has now affected millions of people, including people in France. There are reports in the media about increased stress, anxiety and isolation for the entire population. Likewise, there are many concerns regarding people with mental health issues including people experiencing psychotic symptoms. Thus, studies are needed to understand better the effects of the COVID-19 pandemic and related government measures (e.g., self-isolation) on the mental health and specifically on psychotic experiences. To reach this aim the investigators designed an online survey evaluating people's perceptions of the COVID-19 pandemic and government measures, their habits during the isolation period, to what extent they feel lonely, how they are managing their emotions, their general emotional state and finally the presence of psychotic experiences. Participants will be invited to complete these measures three times. Participants will complete the survey again in 1 week and then in 1 month.

The specific goals of this project are:

* Determine the association between psychotic symptoms (paranoia and hallucinations) and perception of the COVID-19 pandemic and government measures, level of activity, isolation, emotion regulation, cognitive bias and negative affect at Time 1.
* Determine which factors predict psychotic symptoms one week later and one month later.
* Explore changes across time on these measures.

Methodology:

The entire study will be conducted online. Participants will be assessed at baseline_ T1: Peak of the COVID-19 pandemic; T2: 1 week after T1; T3: 1 month after T1.

Participants will provide their informed consent. At these assessment moments, they will complete a set of self-report measures assessing COVID-19 related psychological aspects, emotion regulation, current levels of activity, cognitive bias, as well as paranoid ideation and hallucinatory experiences.

- Participants will create their own ID code (so the investigators can then match their data) and when providing their informed consent to the study they would give us their email addresses so the investigators could contact them to fill out the measures in the 2nd/3rd assessment moment

Sample size:

The investigators have not set a minimum/maximum sample size for this study. The study will remain open until the end of the self-isolation period in France. The investigators hope to recruit at least 600 participants.

List of self-report measures:

* Behavioral activation for Depression Scale
* The UCLA Loneliness Scale
* The Brief Experiential Avoidance Questionnaire
* Cognitive Emotional Regulation Questionnaire
* items measuring cognitive restructuring and catastrophisation
* Repetitive Thinking Questionnaire
* Cognitive bias questionnaire for Psychosis
* Depression Anxiety and Stress Scale
* Paranoia Scale
* Cardiff Anomalous Perceptions Scale

ELIGIBILITY:
Inclusion criteria:

* Individuals from the general population with or without a mental disorder
* French native speaker
* Majority 18 years and more

Exclusion criteria:

* Patient refusing to participate in research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals from the general population with or without a mental disorder
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Total score of the Cardiff Anomalous Perceptions Scale (CAPS) | inclusion, 1 week after inclusion and 1 month after inclusion
  The CAPS is a 32-item self-report scale designed to measure perceptual anomalies and hallucinatory experience that has already been validated in clinical and nonclinical populations. Each of the 32 items involves a question related to a specific hallucinatory experience to which the participant can answer 'yes' or 'no'. If the participant answers 'yes' they are asked to rate how distressing, how intrusive and how often the experience occurs on separate 1-5 rated Likert scales. The scale total is calculated as the total number items responded to with 'yes' (possible range 0-32) and the subscale totals are calculated as the total of the subscale items (possible range 0-160)

SECONDARY OUTCOMES:
Paranoia Scale | inclusion, 1 week after inclusion and 1 month after inclusion
  Paranoia Scale : this self-report scale is widely used in the assessment of paranoia in the general population.
  The scale is comprised of a set of 20 items, answered in a Likert-like scale ranging from 1 (never) to 5 (always). Scores can vary between 20 and 100, where higher scores indicate greater paranoid ideation

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Raffard, PhD, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC